CLINICAL TRIAL: NCT05141422
Title: A Single-centre, Single-arm, Open-label and Fixed-sequence Drug-drug Interaction Study to Evaluate the Effect of Efavirenz on the Pharmacokinetics of SHR2150 in Healthy Chinese Subjects
Brief Title: A Drug-drug Interaction Study of SHR2150 on Healthy Chinese Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR2150-I-105
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Human Immunodeficiency Virus Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a single-centre, single-arm, open-label and fixed-sequence clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR2150+ efavirenz
  Interventions: Drug: SHR2150 tablet、efavirenz

INTERVENTIONS:
Drug: SHR2150 tablet、efavirenz — SHR2150 tablet single dose, Efavirenz single dose.

SUMMARY:
The study is a single-centre, open-label, fixed-sequence, self-controlled clinical trial. It is planned to enroll 20 healthy adult subjects.

Subjects will take SHR2150 on Day 1 and Day 21, and take efavirenz from Day 7 to Day 26.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can communicate well with the researcher, understand and comply with the requirements of this study, and understand and sign the informed consent;
2. Healthy subjects aged 18 ~ 45 (including the boundary value), male and female;
3. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, body mass index (BMI) within the range of 18 ~ 26 kg/m2 (including the boundary value) (BMI= weight (kg)/height 2 (m2));
4. The physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, abdominal B-ultrasound, and chest radiograph are normal or have no clinical significance;
5. The subjects with reproduction ability must agree to take effective contraceptive measures after signing the informed consent form and within 7 months (for female) or 4 months (for male) until the last medication.

Exclusion Criteria:

1. Anyone who has suffered from any clinical serious disease such as the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease which can affect the study results;
2. Those who have undergone surgery within 3 months before the trial, or plan to perform surgery during the study period;
3. Those whose 12-lead ECG is abnormal with clinically significant or ECG QT interval (QTcF) ≥ 450 ms (for male) or > 460 ms (for female) or < 300 ms;
4. Those who donated blood or suffered heavy blood loss (≥400 mL), received blood transfusions, or used blood products within 3 months before enrollment;
5. Have a history of allergies to drugs, food or other substances;
6. Those who have used soft drugs or hard drugs; or those with positive results in urine drug abuse screening;
7. Those who have participated in any clinical trials and have taken study drugs within 3 months before the first administration;
8. Those who have taken any medicine within 1 month before the first administration (including prescription medicines, non-prescription medicines, Chinese herbal medicines, vitamins, calcium tablets and other food supplements), especially the drugs which have any effect on CYP3A4;
9. Regular drinkers within 3 months before the test, that is, drinking more than 15 g of alcohol per day (15 g alcohol = 450 mL of beer, or 50 mL of spirits, or 150 mL of wine), and any alcohol-containing products cannot be stopped during the study;
10. Hepatitis B virus surface antigen is positive, or hepatitis C virus antibody is positive, or treponema pallidum antibody is positive, or human immunodeficiency virus antibody is positive;
11. Women with pregnancy or within lactation period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-22 (Estimated)

PRIMARY OUTCOMES:
Tmax | from Day 1 to Day 7 after the first dose and from Day 21 to Day 27 after the second dose
  Time to maximum observed serum concentration (Tmax) for SHR2150 after Single dose
Cmax | from Day 1 to Day 7 after the first dose and from Day 21 to Day 27 after the second dose
  Maximum observed serum concentration (Cmax) for SHR2150 after Single dose
AUC0-t | from Day 1 to Day 7 after the first dose and from Day 21 to Day 27 after the second dose
  Area under the plasma concentration versus time curve (AUC0-t) for SHR2150 after Single dose
AUC0-inf | from Day 1 to Day 7 after the first dose and from Day 21 to Day 27 after the second dose
  Area under the plasma concentration versus time curve (AUC0-inf ) for SHR2150 after Single dose
T1/2 | from Day 1 to Day 7 after the first dose and from Day 21 to Day 27 after the second dose
  Time to elimination half-life (T1/2) for for SHR2150 after Single dose

SECONDARY OUTCOMES:
Number of subjects with adverse events and the severity of adverse events | from Day 1 to Day 37 after the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- The People's Hospital of Liaoning Province, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided